CLINICAL TRIAL: NCT01550822
Title: HEALS (Healthy Eating And Lifestyle After Stroke): A Pilot Trial of a Multidisciplinary Lifestyle Intervention Program
Brief Title: HEALS (Healthy Eating And Lifestyle After Stroke)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Los Amigos Research and Education Institute (Other)
Collaborators: American Heart Association (Other); University of California, Los Angeles (Other); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 114
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Stroke
Keywords: stroke, lifestyle habits
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HEALS (Active Comparator): Intervention group which will receive group clinics addressing smoking cessation, healthy eating, physical activity, and the risk factors of stroke.
  Interventions: Other: HEALS
- Usual Care (No Intervention): This group will receive usual care for stroke survivors

INTERVENTIONS:
Other: HEALS
  Arms: HEALS

SUMMARY:
This lifestyle intervention plan will improve healthy lifestyle practices (diet, exercise, and smoking cessation) among stroke survivors and result in a reduction in measures of general and abdominal obesity.

DETAILED DESCRIPTION:
Study data collection will consist of a baseline and outcome study visit. Each visit will consist of a survey and physical exam to collect height, weight and body measurements.

Outcome measures include:

1. Physical Activity: Collected via survey using a version of the International Physical Activity Questionnaire
2. Diet: Collected via survey using the Brief Dietary Assessment Tools for Hispanics
3. Body Mass Index (BMI): Collected via physical exam following the Alaska State Department of Health and Social Services BMI Guidelines
4. Abdominal Obesity: Collected via physical exam following the NIH Standard Circumference methods.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Completed 12 month SUSTAIN trial (SUSTAIN criteria: age ≥ 40 years, acute TIA or ischemic stroke within the prior one month and systolic blood pressure (SBP) >120 mm Hg).
* Phase II: Stroke or TIA > 3 months prior to screening date, age > 20 years, blood pressure (SBP) > 120 mm Hg.

Exclusion Criteria:

* Phase I and Phase II: Same as SUSTAIN criteria: medical condition limiting participation in follow up assessments, severe cognitive impairment (MMSE ≤24), and severe global disability (modified Rankin ≥3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Physical activity | 6 months
  90 minutes/week moderate activity; change in minutes of physical activity/week
Diet | 6 months
  ≥5 servings fruits/vegetables/day; change in # servings fruits/vegetables/day
BMI | 6 months
  BMI 18.5-24.9 kg/m2; change in BMI

SECONDARY OUTCOMES:
Abdominal obesity | 6 months
  achieve <88cm for F and <102cm for M; change in waist circumference

CONTACTS AND LOCATIONS:
Locations (1):
- Rancho Los Amigos National Rehabilitation Center, Downey, California, United States

REFERENCES:
- [Derived] Towfighi A, Cheng EM, Hill VA, Barry F, Lee M, Valle NP, Mittman B, Ayala-Rivera M, Moreno L, Espinosa A, Dombish H, Wang D, Ochoa D, Chu A, Atkins M, Vickrey BG. Results of a Pilot Trial of a Lifestyle Intervention for Stroke Survivors: Healthy Eating and Lifestyle after Stroke. J Stroke Cerebrovasc Dis. 2020 Dec;29(12):105323. doi: 10.1016/j.jstrokecerebrovasdis.2020.105323. Epub 2020 Sep 28. PMID 33002791